CLINICAL TRIAL: NCT04243785
Title: A First-In-Human, Open-Label, Escalating Multiple-Dose Study to Evaluate the Safety, Toxicity, and Pharmacokinetics of BTX-A51 Alone and in Combination With Azacitidine in Patients With Relapsed or Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Brief Title: A Study of BTX-A51 in People With Relapsed or Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Edgewood Oncology Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTX-A51-001
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1a (Monotherapy Cohort Escalation) (Experimental): Dosing in this phase of the study consists of the first cycle of therapy (i.e., 28 days consisting of 3 weeks of treatment followed by 1 week with no study drug). The BTX-A51 starting dose for Cohort 1 is 1 mg, to be given 5 days per week (maximum weekly dose of 5 mg). Beginning with Cohort 2, doses are intended to be administered 3 days per week. Barring dose-limiting toxicity (DLT), sequential dose escalation of BTX-A51 is planned with up to a total of eight dose levels to a maximum of 21 mg (63 mg/week); on the basis of these an MTD will be identified. The numbers of participants and actual doses administered will be determined using a Bayesian optimal interval (BOIN) design to determine the DLTs and MTD of BTX-A51.
  Interventions: Drug: BTX-A51
- Part 1b (Monotherapy Cohort Expansion) (Experimental): Dosing in this phase of the study consists of the first cycle of therapy (i.e., 28 days consisting of 3 weeks of treatment followed by 1 week with no study drug). Part 1b will continue at the MTD or the highest dose achieved in Phase 1a.
  Interventions: Drug: BTX-A51
- Part 1c (Azacitidine Combination Dose Escalation) (Experimental): After determination of MTD and RP2D from Part 1a, combination dose escalation in Part 1c may begin. Patients with AML will receive BTX-A51 combined with azacitidine in escalating BTX-A51 dose cohorts. Dosing in this stage of the study consists of the first cycle of therapy (i.e., 28 days). The starting dose of BTX-A51 will be RP2D. Part 1c will follow a BOIN design as described for Part 1a. The numbers of patients and actual doses administered will be determined in response to DLTs a. There will be at least 3 patients per cohort.
  Interventions: Drug: BTX-A51; Drug: Azacitidine

INTERVENTIONS:
Drug: BTX-A51 — Orally administered capsules available in strengths of 0.5 mg, 1.0 mg, 2.0 mg and 7 mg.
Drug: Azacitidine — Azacitidine will be administered IV or SC 75 mg/m2 QD on Days 1-7 of each 28-day cycle.
  Arms: Part 1c (Azacitidine Combination Dose Escalation)

SUMMARY:
This is an open-label, dose escalation study to evaluate the safety, toxicity, and pharmacokinetics (PK) as well as preliminary efficacy of BTX-A51 capsules in participants with relapsed or refractory acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS).

The study will be done in three parts. Part 1a (Monotherapy Dose Escalation) of this study is designed to determine the dose-limiting toxicities (DLTs) and maximum tolerated dose (MTD) of orally administered BTX-A51 in up to 35 participants who are evaluable for toxicity. Once the MTD is determined, it is planned that an additional 15 participants will be enrolled in Part 1b (Monotherapy Cohort Expansion) of this study for additional experience with safety and efficacy, and to determine the recommended Phase 2 dose (RP2D) which may or may not be different from the MTD. After determination of MTD and RP2D from Part 1a, Part 1c (Azacitidine Combination Dose Escalation) will enroll up to 30 participants.

Continued treatment will be available under this study protocol for up to eight 28-day cycles (Continued Treatment Phase) if the Investigator judges the benefit outweighs the risk.

Once BTX-A51 treatment has completed, participants will be contacted by telephone every 3 months for up to 2 years after their last treatment for survival status and anticancer therapy (Overall Survival Follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Demonstration of understanding and voluntarily signing of an informed consent form
* Age ≥ 18 years
* Diagnosis of acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) according to the World Health Organization classification and, with respect to MDS, that is high risk; participants must have refractory or relapsed disease and be ineligible for or have exhausted standard therapeutic options that would otherwise be likely to provide clinical benefit
* Eastern Cooperative Oncology Group performance status ≤ 2 and life expectancy of ≥ 6 weeks
* Adequate organ function (Grade 1 serum creatinine; Grade 1 total bilirubin; aspartate aminotransferase and/or alanine transaminase ≤ 2 × ULN)
* Females of childbearing age must not be pregnant at time of Screening/beginning of treatment and agree to either abstain from sexual intercourse or use highly effective methods of contraception (for up to 3 months after last dose of study drug)
* Males sexually active with a woman of childbearing age must agree to use barrier method of birth control during and after the study (up to 3 months after last dose of study drug)

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* White blood cell count > 20 x 10^9/L
* Receipt of cancer chemotherapy (other than hydroxyurea) within 2 weeks prior to the start of study drug
* In participants who have undergone autologous or allogeneic stem cell transplantation: transplantation within the 3 months prior to Screening; active graft-versus-host disease requiring anything other than topical corticosteroids and budesonide; treatment with systemic immunosuppressive medications including high-dose steroids (≥ 20 mg prednisolone or equivalent per day), or calcineurin inhibitors (e.g., cyclosporine, tacrolimus) for at least 1 week prior to Screening, and sirolimus, mycophenylate mofetil, azathioprine, or ruxolitinib for at least 2 weeks prior to Screening
* Immediate life-threatening severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Persistent toxicities from prior treatment of Grade 2 or higher
* Active uncontrolled systemic fungal, bacterial, mycobacterial, or viral infection
* Clinically significant cardiac disease
* Known dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Any other concurrent medical condition or disease that is likely to interfere with study procedures or results, or that, in the opinion of the Investigator, would constitute a hazard for participating in this study
* If female, pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-06 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | Up to a total of eight 28-day cycles (approximately 224 days)
  A DLT is defined as a severe or clinically significant adverse event (AE) or abnormal laboratory value (Grade 3 or greater, unless otherwise specified) starting with the first dose on Cycle 1 Day 1, unless it is clearly related to disease progression, intercurrent illness, preexisting condition, or concomitant medications. DLTs are based on National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Number of participants with non-serious AEs and serious AEs (SAEs) | Up to a total of eight 28-day cycles (approximately 224 days)
  The severity/intensity of AEs will be graded based upon the participant's symptoms according to the NCI CTCAE Version 5.0
Number of participants with laboratory abnormalities and/or AEs | Up to a total of eight 28-day cycles (approximately 224 days)
  Number of participants with potentially clinically significant laboratory values; toxicity will be graded and reported according to the NCI CTCAE Version 5.0
Number of participants with 12-lead electrocardiogram (ECG) abnormalities and/or AEs | Up to a total of eight 28-day cycles (approximately 224 days)
  Number of participants with potentially clinically significant 12-lead ECG findings; toxicity will be graded and reported according to the NCI CTCAE Version 5.0
Number of participants with echocardiogram (ECHO) abnormalities and/or AEs | Up to a total of eight 28-day cycles (approximately 224 days)
  Number of participants with potentially clinically significant ECHO abnormalities and/or AEs, such as elevated or abnormal left ventricular ejection fraction (LVEF) or abnormal Global Longitudinal Strain (GLS)
Number of participants with vital sign abnormalities and/or AEs | Up to a total of eight 28-day cycles (approximately 224 days)
  Number of participants with potentially clinically significant vital sign values; toxicity will be graded and reported according to the NCI CTCAE Version 5.0
Number of participants with physical examination abnormalities and/or AEs | Up to a total of eight 28-day cycles (approximately 224 days)
  Number of participants with potentially clinically significant physical examination findings; toxicity will be graded and reported according to the NCI CTCAE Version 5.0
Maximum tolerated dose (MTD) | Up to 28 days (one cycle) for each dosing cohort in Phase 1a
  The DLTs are to be evaluated for determination of the MTD. The MTD will be the dose for which the isotonic estimate of the toxicity rate is closest to the target toxicity rate of 0.3. If there are ties, the higher dose level when the isotonic estimate is lower than the target toxicity rate will be identified and the lower dose level selected when the isotonic estimate is greater than or equal to the target toxicity rate.
Recommended Phase 2 dose (RP2D) | Up to 28 days (one cycle) for each dosing cohort in Phase 1b
  The DLTs are to be evaluated based on cumulative safety/PK data in participants treated in Phase 1b for determination of the RP2D (which may or may not differ from the MTD)

SECONDARY OUTCOMES:
Complete remission (CR) for participants with acute myeloid leukemia (AML) | Up to a total of eight 28-day cycles (approximately 224 days)
  CR is defined as free of all symptoms related to leukemia and with an absolute neutrophil count (ANC) ≥ 1.0 × 10^9/L (1000/µL), platelet count ≥ 100 × 10^9/L (100,000/µL), and normal bone marrow (BM) with < 5 percent blasts; absence of circulating blasts and blasts with Auer rods
Complete remission with incomplete blood count recovery (CRi) for participants with AML | Up to a total of eight 28-day cycles (approximately 224 days)
  CRi is defined as all CR criteria except for residual neutropenia (ANC < 1.0 × 10^9/L [1000/µL]) or thrombocytopenia (platelet count < 100 × 10^9/L [100,000/µL])
Morphologic leukemia-free state (MLFS) for participants with AML | Up to a total of eight 28-day cycles (approximately 224 days)
  MLFS is defined as BM blasts < 5 percent; absence of blasts with Auer rods; absence of extramedullary disease; no hematologic recovery required. Marrow should not barely be "aplastic;" at least 200 cells should be enumerated or cellularity should be at least 10 percent.
Partial remission (PR) for participants with AML | Up to a total of eight 28-day cycles (approximately 224 days)
  PR is defined as all hematologic criteria of CR; decrease of BM blast percentage to 5 - 25 percent; and decrease of pretreatment BM blast percentage by at least 50 percent
Complete remission (CR) for participants with high-risk myelodysplastic syndrome (MDS) | Up to a total of eight 28-day cycles (approximately 224 days)
  CR is defined as free of all symptoms related to leukemia and with an ANC ≥ 1.0 × 10^9/L, platelet count ≥ 100 × 10^9/L, BM ≤ 5 percent myeloblasts, with normal maturation of all cell lines, hemoglobin ≥ 11 g/dL, and no blasts in peripheral blood (PB)
Partial remission (PR) for participants with high-risk MDS | Up to a total of eight 28-day cycles (approximately 224 days)
  PR is defined as all CR criteria with ≥ 50 percent decrease in BM blasts over pre-treatment (but still > 5 percent)
Hematologic improvement (HI) for participants with high-risk MDS | Up to a total of eight 28-day cycles (approximately 224 days)
  The International Working Group criteria for HI defining specific responses of cytopenias in the three hematopoietic lineages: erythroid (HI-E), platelet (HI-P), and neutrophil (HI-N)
Overall survival and event-free survival in participants with AML or high-risk MDS | Up to 2 years after participant's last dose of BTX-A51 or upon death, whichever occurs first
  Follow-up will occur by telephone contact once every 3 months for assessment of survival status and bone marrow transplant (BMT) conditioning or other new antineoplastic therapies since discontinuation of study drug; the cause of death will be documented. Disease assessment will be collected for participants who discontinue study medication due to any reason other than progression or death. If a participant has not progressed or died, progression-free survival is censored at the date of last follow up. The distribution of time-to-event endpoints will be estimated using the method of Kaplan and Meier.
PK parameter: Maximum observed plasma concentration (Cmax) | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Maximum observed plasma drug concentration after the first dose
PK parameter: Time of maximum plasma concentration (Tmax) | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Time to reach Cmax
PK parameter: Plasma CmaxD5 | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Maximum observed plasma drug concentration after the dose on Day 5
PK parameter: Plasma TmaxD5 | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Time to reach CmaxD5
PK parameter: C0 | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Pre-dose concentrations in PK blood samples on dosing days
PK parameter: AUC0-24 | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Area under the curve from time 0 to 24 hours after the first dose
PK parameter: AUC0-24D5 | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  AUC from time 0 to 24 hours after the dose on Day 5
PK parameter: Terminal elimination rate constant (Kel) | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Calculated by linear least-squares regression analysis from a semi-log plot of the plasma concentration versus time curve after the Day 5 dose
PK parameter: Terminal elimination phase half-life (t1/2) | During Cycle 1 for each dosing cohort in Phase 1a on Days 1, 3, and 5 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose); Days 2, 4, 6, 7, 8; and Day 15 (pre-dose and approximately 1, 2, 3, 5, 8, and 12 hours post-dose)
  Estimated after the Day 5 dose, calculated as 0.693/Kel

CONTACTS AND LOCATIONS:
Overall Officials: Zung Thai, MD, Study Director — Edgewood Oncology Inc.
Locations (3):
- United States (3):
  - City of Hope National Medical Center, Duarte, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas